CLINICAL TRIAL: NCT04926246
Title: Formulation Selection and Subsequent Optimization of Oral Formulations of BI 685509 in Healthy Male Subjects (Open-label, Randomized, Single-dose Design Study in up to Three Parts; Trial Part 1: Five-period Crossover; Optional Trial Parts 2 & 3: Fourperiod Crossover)
Brief Title: A Study in Healthy Men to Find the Best Formulation of BI 685509 and to Test How it is Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1366-0024
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Study in up to three parts:
  Trial part 1: five-period crossover Optional trial part 2: four-period crossover Optional trial part 3: four-period crossover
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1: R1-T2-T4-T1-T3 (Experimental)
  Interventions: Drug: R1: Reference Product X; Drug: T1: Test Product M; Drug: T2: Test Product N; Drug: T3: Test Product O; Drug: T4: Test Product O
- Part 1: T1-T4-T2-T3-R1 (Experimental)
  Interventions: Drug: R1: Reference Product X; Drug: T1: Test Product M; Drug: T2: Test Product N; Drug: T3: Test Product O; Drug: T4: Test Product O
- Part 1: T2-T1-T3-R1-T4 (Experimental)
  Interventions: Drug: R1: Reference Product X; Drug: T1: Test Product M; Drug: T2: Test Product N; Drug: T3: Test Product O; Drug: T4: Test Product O
- Part 1: T3-R1-T1-T4-T2 (Experimental)
  Interventions: Drug: R1: Reference Product X; Drug: T1: Test Product M; Drug: T2: Test Product N; Drug: T3: Test Product O; Drug: T4: Test Product O
- Part 1: T4-T3-R1-T2-T1 (Experimental)
  Interventions: Drug: R1: Reference Product X; Drug: T1: Test Product M; Drug: T2: Test Product N; Drug: T3: Test Product O; Drug: T4: Test Product O
- Part 2: R2-T7-T6-T5 (Experimental)
  Interventions: Drug: R2: Reference Product Y; Drug: T5: Test Product P; Drug: T6: Test Product P; Drug: T7: Test Product Q
- Part 2: T5-T6-T7-R2 (Experimental)
  Interventions: Drug: R2: Reference Product Y; Drug: T5: Test Product P; Drug: T6: Test Product P; Drug: T7: Test Product Q
- Part 2: T6-T5-R2-T7 (Experimental)
  Interventions: Drug: R2: Reference Product Y; Drug: T5: Test Product P; Drug: T6: Test Product P; Drug: T7: Test Product Q
- Part 2: T7-R2-T5-T6 (Experimental)
  Interventions: Drug: R2: Reference Product Y; Drug: T5: Test Product P; Drug: T6: Test Product P; Drug: T7: Test Product Q
- Part 3: R3-T10-T9-T8 (Experimental)
  Interventions: Drug: R3: Reference Product Z; Drug: T8: Test Product S; Drug: T9: Test Product S; Drug: T10: Test Product U
- Part 3: T8-T9-T10-R3 (Experimental)
  Interventions: Drug: R3: Reference Product Z; Drug: T8: Test Product S; Drug: T9: Test Product S; Drug: T10: Test Product U
- Part 3: T9-T8-R3-T10 (Experimental)
  Interventions: Drug: R3: Reference Product Z; Drug: T8: Test Product S; Drug: T9: Test Product S; Drug: T10: Test Product U
- Part 3: T10-R3-T8-T9 (Experimental)
  Interventions: Drug: R3: Reference Product Z; Drug: T8: Test Product S; Drug: T9: Test Product S; Drug: T10: Test Product U

INTERVENTIONS:
Drug: R1: Reference Product X — under fasted conditions
  Arms: Part 1: R1-T2-T4-T1-T3; Part 1: T1-T4-T2-T3-R1; Part 1: T2-T1-T3-R1-T4; Part 1: T3-R1-T1-T4-T2; Part 1: T4-T3-R1-T2-T1
Drug: T1: Test Product M — under fasted conditions
  Arms: Part 1: R1-T2-T4-T1-T3; Part 1: T1-T4-T2-T3-R1; Part 1: T2-T1-T3-R1-T4; Part 1: T3-R1-T1-T4-T2; Part 1: T4-T3-R1-T2-T1
Drug: T2: Test Product N — under fasted conditions
  Arms: Part 1: R1-T2-T4-T1-T3; Part 1: T1-T4-T2-T3-R1; Part 1: T2-T1-T3-R1-T4; Part 1: T3-R1-T1-T4-T2; Part 1: T4-T3-R1-T2-T1
Drug: T3: Test Product O — under fasted conditions
  Arms: Part 1: R1-T2-T4-T1-T3; Part 1: T1-T4-T2-T3-R1; Part 1: T2-T1-T3-R1-T4; Part 1: T3-R1-T1-T4-T2; Part 1: T4-T3-R1-T2-T1
Drug: T4: Test Product O — under fed conditions
  Arms: Part 1: R1-T2-T4-T1-T3; Part 1: T1-T4-T2-T3-R1; Part 1: T2-T1-T3-R1-T4; Part 1: T3-R1-T1-T4-T2; Part 1: T4-T3-R1-T2-T1
Drug: R2: Reference Product Y — under fasted conditions
  Arms: Part 2: R2-T7-T6-T5; Part 2: T5-T6-T7-R2; Part 2: T6-T5-R2-T7; Part 2: T7-R2-T5-T6
Drug: T5: Test Product P — under fasted conditions
  Arms: Part 2: R2-T7-T6-T5; Part 2: T5-T6-T7-R2; Part 2: T6-T5-R2-T7; Part 2: T7-R2-T5-T6
Drug: T6: Test Product P — under fed conditions
  Arms: Part 2: R2-T7-T6-T5; Part 2: T5-T6-T7-R2; Part 2: T6-T5-R2-T7; Part 2: T7-R2-T5-T6
Drug: T7: Test Product Q — under fasted conditions
  Arms: Part 2: R2-T7-T6-T5; Part 2: T5-T6-T7-R2; Part 2: T6-T5-R2-T7; Part 2: T7-R2-T5-T6
Drug: R3: Reference Product Z — under fasted conditions
  Arms: Part 3: R3-T10-T9-T8; Part 3: T10-R3-T8-T9; Part 3: T8-T9-T10-R3; Part 3: T9-T8-R3-T10
Drug: T8: Test Product S — under fasted conditions
  Arms: Part 3: R3-T10-T9-T8; Part 3: T10-R3-T8-T9; Part 3: T8-T9-T10-R3; Part 3: T9-T8-R3-T10
Drug: T9: Test Product S — under fed conditions
  Arms: Part 3: R3-T10-T9-T8; Part 3: T10-R3-T8-T9; Part 3: T8-T9-T10-R3; Part 3: T9-T8-R3-T10
Drug: T10: Test Product U — under fasted conditions
  Arms: Part 3: R3-T10-T9-T8; Part 3: T10-R3-T8-T9; Part 3: T8-T9-T10-R3; Part 3: T9-T8-R3-T10

SUMMARY:
The main objective of this trial is to select a formulation and to optimize the identified formulation of BI 685509, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive) at the time of signing informed consent
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive) at the time of signing informed consent
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who are sexually active must use with their partner, highly effective contraception from the time of administration of trial medication until 30 days after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
  * Condoms plus surgically sterilised partner (including hysterectomy) or
  * Condoms plus intrauterine device or
  * Condoms plus partner of non-childbearing potential (including homosexual men) Subjects are required to use condoms to prevent unintended exposure of the partner (both, male and female) to the study drug via seminal fluid. Male subjects should use a condom throughout the study and for 30 days after last Investigational Medicinal Product (IMP) administration. Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active with their partner, they must comply with the contraceptive requirements detailed above.

Male subjects should not donate sperm for the duration of the study and for at least 30 days after last IMP administration.

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 60 to 90 mmHg, or pulse rate outside the range of 40 to 100 bpm at screening and pre-dose of first period
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator, including not resolved post-vaccination reactions
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, dermatological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair, unless within the last 12 months)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 685509 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 5 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 685509 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com